CLINICAL TRIAL: NCT02544659
Title: Unrandomized, Open Label Single-center Study to Assess the Long Term Efficacy of Intravenous Bisphosphonates for Bone Marrow Edema in Patients With SAPHO Syndrome
Brief Title: Efficacy of Bisphosphonates in Patients With Synovitis, Acne, Pustulosis, Hyperostosis, and Osteitis (SAPHO) Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-SAPHO-01
Record Dates: First submitted 2015-08-28; First posted 2015-09-09 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2015-09

CONDITIONS: SAPHO Syndrome
Keywords: Treatment; Bisphosphonates; Response rate
MeSH Terms: conditions — Acquired Hyperostosis Syndrome | interventions — Pamidronate

ARMS (1):
- pamidronate disodium (Experimental): the patients will be administered intravenous pamidronate disodium
  Interventions: Drug: pamidronate disodium

INTERVENTIONS:
Drug: pamidronate disodium — the patients will be administered pamidronate disodium 1 mg/kg, IV, QD, for 3 days, and every 3 month (up to month 6)

SUMMARY:
This study is designed to evaluate long term efficacy of intravenous bisphosphonates for bone marrow edema in patients with SAPHO syndrome.

DETAILED DESCRIPTION:
The study will evaluate the long term efficacy at 3 days, 3 and 6 months after pamidronate disodium administered. Patients will be administered pamidronate disodium 1 mg/kg, IV, QD, for 3 days, and every 3 months (up to month 6).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 and 70 years
2. Only 1 of the 4 inclusion criteria is sufficient to arrive at a diagnosis of SAPHO syndrome：

   * Osteo-articular manifestations of acne conglobata, acne fulminans, or hidradenitis suppurativa
   * Osteo-articular manifestations of PPP
   * Hyperostosis (of the anterior chest wall, limbs or spine) with or without dermatosis
   * CRMO involving the axial or peripheral skeleton with or without dermatosis Palmoplantar pustulosis(PPP); chronic recurrent multifocal osteomyelitis(CRMO)
3. MRI shows bone marrow edema in affected site in patients
4. Blood serum of patients show the normal white blood cell count, liver and renal function
5. Patients who like to be followed up for 1 years
6. Other protocol defined inclusion criteria may apply

Exclusion Criteria:

1. Women in pregnancy or lactation.
2. Septic osteomyelitis
3. Infectious chest wall arthritis
4. Infections PPP
5. Palmo-plantar keratodermia
6. DISH except for fortuitous association
7. Osteoarticular manifestations of retinoid therapy
8. Other protocol defined exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
response to the treatment by the change of MRI result at screening, baseline, month 3 and month 6 | 3 and 6 month (up to 6 month)

SECONDARY OUTCOMES:
physician's global assessment of disease activity at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of Visual Analogue ale/Score (VAS) at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of bath ankylosing spondylitis disease activity index (BASDAI) at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of bath ankylosing spondylitis functional index (BASFI) at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of bath ankylosing spondylitis metroloty index (BASMI) at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of ankylosing spondylitis disease activity score (ASDAS) at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of erythrocyte sedimentation rate (ESR) at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of high sensitivity-C reaction protein (hs-CRP) at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of Osteocalcin at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)
response to the treatment by the change of beta-Crosslaps (beta-CTx) at screening, baseline, month 3 and month 6 | 3 days, 3 and 6 month (up to 6 month)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Li, Master, Principal Investigator — Department of Traditional Chinese Medicine, Peking Union Medical College Hospital